CLINICAL TRIAL: NCT00787592
Title: A Prospective Comparison of Silver Sulfadiazine Cream and Collagenase Ointment for the Treatment of Burns in Children
Brief Title: SSD vs Collagenase in Pediatric Burn Patients
Status: Completed | Type: Observational
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Sponsor
Other Study IDs: 07-11-174
Record Dates: First submitted 2008-11-06; First posted 2008-11-07 (Estimated); Last update posted 2021-01-08 (Actual); Status verified 2021-01

CONDITIONS: Burns
Keywords: Burns; children; collagenase; silver sulfadiazine; Childhood burns
MeSH Terms: conditions — Burns

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Silver Sulfadiazide (SSD): Patients that receive SSD as the topical debriding agent
- Collagenase: Patients that receive collagenase as the debriding agent

SUMMARY:
The objective of this study is to evaluate the outcomes of children with burn injury with regard to the utilization of Silver sulfadiazine (SSD) cream and Collagenase ointment. The primary outcome variable will be need for skin grafting. The specific aim of the study is to prospectively collect data to determine if SSD is superior to Collagenase with regard to avoiding the need for skin grafting.

DETAILED DESCRIPTION:
During the treatment of burns, the wounds must be repeatedly debrided to remove loose and adherent dead tissue (eschar) until it is determined that the wound will require skin grafting for coverage or that the wound will re-epithelialize. The eschar associated with burn injury eventually will separate from the burn bed through proteolytic enzymes that are produced naturally in the skin or by colonizing bacteria. During this acute treatment timeframe, agents are used that can help with removal of the eschar. SSD is an antimicrobial agent that sterilizes the wound, thus preventing infection and allowing the natural proteolytic enzymes in the skin to act on the eschar leading to separation during the mechanical debridement treatment regimen. SSD was initially introduced in the 1960's and has been a mainstay of treatment for the care of burns since. It is currently used in the CMH burn unit.

Collagen is a protein that is highly present in skin (~75% of dry weight of skin), and is the dominant protein that must be divided to allow for eschar separation. Collagenase is an exogenous enzyme that breaks down native and denatured collagen. Collagenase will not however breakdown healthy, normal collagen. Collagenase is FDA approved for the treatment of burns and is now used by many burn units including the burn unit at CMH. Currently, in this institution, both SSD and collagenase are being used for the removal of eschar. Unfortunately, there has not been a properly performed prospective randomized comparison of these two regimens in children, despite the widespread use of both regimens. Because of the uncertain data regarding these approaches, as well as the fact that we currently perform both approaches here, we feel that there is equipoise in regard to the techniques. We plan to perform a prospective randomized trial comparing SSD and Collagenase in children that sustain burns and are admitted to CMH for debridement of their burns. We have reviewed our historical experience using collagenase and SSD. Utilizing the need for skin graft rates from this historical population, a sample size of 75 patients in each arm has been calculated. This sample size calculation was performed using a standard alpha and beta of 0.05 and 0.8, respectively, and assumes a 10% attrition rate. The primary endpoint for this study will be the need for skin grafting in children that sustain a burn of sufficient depth to require admission and debridement of eschar.

ELIGIBILITY:
Inclusion Criteria:

1. Partial thickness burn
2. Less than 25% total body surface area burn
3. Less than 18 years of age
4. Greater than 2 months of age

Exclusion Criteria:

1. Greater than 25% total body surface burn
2. 18 years of age or older
3. Younger than 2 months of age
4. Allergy to sulfa

Ages: 2 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children between the ages of 2 months and 18 years of age that have at least second degree burns that involve less than 25% of their total body surface area.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2008-01 (Actual); Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Need for skin grafting | 10 days

SECONDARY OUTCOMES:
Development of burn contractures | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J Ostlie, MD, Principal Investigator — Children's Mercy Hospital and Clinics
Locations (1):
- Children's Mercy Hospital and Clinics, Kansas City, Missouri, United States

REFERENCES:
- [Background] Hansbrough JF, Achauer B, Dawson J, Himel H, Luterman A, Slater H, Levenson S, Salzberg CA, Hansbrough WB, Dore C. Wound healing in partial-thickness burn wounds treated with collagenase ointment versus silver sulfadiazine cream. J Burn Care Rehabil. 1995 May-Jun;16(3 Pt 1):241-7. doi: 10.1097/00004630-199505000-00004. PMID 7673302
- [Background] Ozcan C, Ergun O, Celik A, Corduk N, Ozok G. Enzymatic debridement of burn wound with collagenase in children with partial-thickness burns. Burns. 2002 Dec;28(8):791-4. doi: 10.1016/s0305-4179(02)00191-2. PMID 12464480
- [Background] Atiyeh BS, Costagliola M, Hayek SN, Dibo SA. Effect of silver on burn wound infection control and healing: review of the literature. Burns. 2007 Mar;33(2):139-48. doi: 10.1016/j.burns.2006.06.010. Epub 2006 Nov 29. PMID 17137719